CLINICAL TRIAL: NCT03008798
Title: Prevention for the Restenosis of Intracranial Artery Stent Implantation Treated With Herbal Medicine C117--PRISIT Trial
Brief Title: Prevention for the Restenosis of Intracranial Artery Stent Implantation Treated With Herbal Medicine C117
Acronym: PRISIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Liaocheng People's Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, jianwen guo, MD, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014A020221074
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Occlusion and Stenosis of Unspecified Cerebral Artery
Keywords: Intracranial Artery; in-stent restenosis; Herbal Medicine
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herbal Medicine C-117 (Experimental): Herbal Medicine C-117 6g granules by mouth,every 12 hours for 1 year
  Interventions: Drug: Herbal Medicine C-117
- The Placebo of Herbal Medicine C-117 (Placebo Comparator): The Placebo of Herbal Medicine C-117 6g granules by mouth,every 12 hours for 1 year
  Interventions: Drug: The Placebo of Herbal Medicine C-117

INTERVENTIONS:
Drug: Herbal Medicine C-117 — C117 formula including 2 herbals and 2 insects
  Arms: Herbal Medicine C-117
Drug: The Placebo of Herbal Medicine C-117
  Arms: The Placebo of Herbal Medicine C-117

SUMMARY:
Prevention for the Restenosis of Intracranial artery Stent Implantation Treated with herbal medicine C117--PRISIT Trial

DETAILED DESCRIPTION:
Intracranial artery stenosis (ICAS) is a common cause of ischemic stroke worldwide. At present, percutaneous transluminal angioplasty and stenting serve as a possible treatment option for ICAS patients, however, intracranial in-stent restenosis(ISR) limited its use in clinical practice, which led to recurrent stroke even death, meanwhile, From the point of chinese medicine, in-stent restenosis(ISR) regard as the unhealthy environmental influences with shapes, therefore, we have design two control group on the basis of conventional secondary prevention, one use herbal medicine for blood-acting and stasis-dissolving, and another use the similar looking placebos, after 12 months of treatment, we will evaluate the rate of all-cause stroke and all-cause mortality, moreover, we also record the Vascular restenosis rate which may cause recurrent ischemic stroke, the aim of this study was to evaluate the safety and efficacy of herbal medicine C-117.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age
2. 70-90% stenosis of intracranial responsible angiopathic area under the DSA angiography (as judged through the WASID method);after operation vascular stenosis less than 50%.
3. The score of mRS≤3
4. To rule out intracranial hemorrhage by CT orMRI
5. Adhere to the medication

Exclusion Criteria：

1. Together with intracranial tumors or AVM
2. The lesion area where implant stent previons
3. Fetch intracranial artery thrombus by emergency surgical operation
4. Vascular serious circuity
5. Myocardial infarction need to antithrombotic
6. MoyaMoya disease or cerebral vasculitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the total number of all-cause mortality and all-cause stroke within 12 months | After 12 months follow-up
  After drug-use 12 months,observe all-cause mortality and all-cause stroke（hemorrhage or ischemic）.

SECONDARY OUTCOMES:
The rate of intracranial in-stent restenosis | After 12 months follow-up period,record the rate of intracranial in-stent restenosis
  After drug-use 12 months,observe the rate of intracranial in-stent restenosis where stent implantation.throgh the test of TCD, digital subtraction angiography.
The complications of intracranial in-stent restenosis | After 12 months follow-up period,record the complications of intracranial in-stent restenosis
  After drug-use 12 months,observe the complications of intracranial in-stent restenosis,including TIA and stroke,even death.
NIH Stroke Scale （NIHSS） | After 12 months follow-up period
  At the time of 6 and 12 months,we will have a follow-up to assess the patient's NIHSS
Bathel index | After 12 months follow-up period
  At the time of 6 and 12 months,we will have a follow-up to assess the patient's NIHSS, Bathel index
modified RANKIN score. | After 12 months follow-up period
  modified RANKIN score.

CONTACTS AND LOCATIONS:
Overall Officials: Yingguang Zhang, MD, Principal Investigator — Guangdong Province Hospital of Tradtional Chinese Medicine; Zhangyong Xia, MD, Principal Investigator — Liaocheng People's Hospital; Jian Yang, MD, Principal Investigator — Liaoning Cancer Hospital & Institute; Wentong Ling, MD, Principal Investigator — Zhangshan People's Hospital